CLINICAL TRIAL: NCT04059640
Title: PMCF Study to Evaluate the Safety and Performance of LiquiBand FIX8® Open Hernia Mesh Fixation Device
Brief Title: PMCF Study of LiquiBand FIX8® OHMF Device
Acronym: LBF8-Open
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: Imarc Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHMF-001
Record Dates: First submitted 2019-08-09; First posted 2019-08-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-01

CONDITIONS: Inguinal Hernia
Keywords: Inguinal Hernia; Mesh Fixation; Surgical Site Wound Closure
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LiquiBand FIX8® OHMF Device (Experimental): Subjects will undergo hernia mesh fixation and topical wound closure using the LiquiBand FIX8® OHMF device.
  Interventions: Device: LiquiBand FIX8 Open Hernia Mesh Fixation Device

INTERVENTIONS:
Device: LiquiBand FIX8 Open Hernia Mesh Fixation Device — Subjects will undergo hernia mesh fixation and topical wound closure using the LiquiBand FIX8® OHMF device.
  Subjects will be evaluated intra-operatively, post-operatively, at discharge, and at 12 months post-operatively. The Liquiband surgical study device is considered a permanent implant.

SUMMARY:
Study to evaluate the safety and performance of LiquiBand FIX8® Open Hernia Mesh Fixation Device.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand and give informed consent to take part in the study
* Subject has a primary inguinal hernia.
* Subject is scheduled to undergo open inguinal hernia repair using the LiquiBand FIX8® OHMF device.
* Subject is willing and able to comply with the protocol assessments at time of surgery and during the post-surgical follow-up period.

Exclusion Criteria:

* Subject is undergoing open repair surgery for recurrent hernia, where the primary surgery was also open. Subjects with recurrent hernia whose primary surgery was laparoscopic are not excluded.
* Subject has an anatomical defect or had prior surgical procedures that in the opinion of the investigator makes them unsuitable for open hernia repair with the LiquiBand FIX8® OHMF device.
* Subject is known to be non-compliant with medical treatment.
* Subject is pregnant or actively breastfeeding.
* Subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study.
* Subject has a known sensitivity to cyanoacrylate or formaldehyde, D&C Violet No.2 dye or any other component of LiquiBand FIX8® OHMF device.
* The hernia mesh to be used in the repair is constructed from Polytetrafluoroethylene (PTFE) or absorbable materials.
* The hernia mesh to be used in the repair is a self-gripping mesh (e.g. ProGrip).
* Subject has active or potential infection at the surgical site.
* Subject has a history of keloid formation.
* Subject has a known vitamin C or zinc deficiency.
* Subject has a connective tissue disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the LiquiBand FIX8 OHMF device | Time of surgery
  Effectiveness will be defined as successful fixation of the hernia mesh (ie not requiring additional fixation by an alternate device) using the LiquiBand FIX8 device at the time of surgery. Based on data pooled from published studies of a similar device (which employs the same cyanoacrylate glue to fix hernia mesh, via a laparoscopic rather than open surgical approach), there has been an observed failure rate of 0.8% in mesh fixation. This study aims to demonstrate non-inferiority of the LiquiBand FIX8 device to a failure rate of 5% (medically acceptable inference).

SECONDARY OUTCOMES:
Safety of the LiquiBand FIX8 OHMF device | 0 (intra-operatively), up to 2 days (discharge from hospital) and 12-months post surgery
  The incidence of adverse events (whether or not determined to be related to the LiquiBand FIX8 Device) will be recorded. Complications assessed during the study will include:
  * Haematoma
  * Seroma
  * Testicular ischaemia and atrophy
  * Surgical site or wound infection/dehiscence
  * Mesh infection
  * Chronic post-operative pain (lasting ≥ 12 months post-surgery
Effectiveness of the LiquiBandFIX8 OHMF device for topical wound closure | Time of surgery
  Defined as successful closure of the incision site using the LiquiBand FIX8 Device (not requiring additional fixation by an alternate device).
Assessment of chronic post-operative pain using the Visual Analogue Scale: the minimal clinically important difference and patient acceptable symptom state. | 12-months post-surgery
  Chronic post-operative pain will be assessed using the following measures:
  * Improvement in post-operative pain from baseline to 12 months post-surgery as measured by the Visual Analogue Scale (0 = no pain to 10 = most pain imaginable); and
  * Analgesic requirements in the 12 months post-surgery
Long term performance of the study device | 12-months post surgery
  Long-term performance will be assessed by rate of hernia recurrence.
Comparison of cost-effectiveness of patients treated with the LiquiBand FIX8 OHMF device compared with costs for those treated using standard surgical technique. | 12-months
  A study-specific outcome model will be used, which will calculate an incremental cost effectiveness ratio (ICER) in terms of quality-adjusted life years (QALYs) achieved with the introduction of the LiquiBand FIX8 OHMF device compared with using a standard surgical technique (suture fixation).
Comparison of costs of patients' clinical events treated with the LiquiBand FIX8 OHMF device compared with costs for those treated using standard surgical technique. | 12-months
  A study-specific outcome model will be used which will calculate an incremental cost effectiveness ratio (ICER) given in terms of clinical events avoided achieved with the introduction of the LiquiBand FIX8 OHMF device compared with using a standard surgical technique (suture fixation).
Clinician satisfaction | 0 (Post Surgery) and upto 2 days (hospital discharge)
  Users will be asked to rate the device on factors relating to ease of use and satisfaction, compared with their experience of other hernia mesh fixation devices. Satisfaction will be assessed using a Likert-type scale (e.g. Very satisfied (1), Satisfied (2), Neither (3), Dissatisfied (4), Very dissatisfied (5))

OTHER OUTCOMES:
Cosmesis of wound closure using the Visual Analogue Scale | 12-months
  Cosmesis of the wound closure will be assessed by the investigator and patient, and measured by Visual Analogue Scale (0 = Very poor cosmetic outcome; to 10 = very good cosmetic outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Mihailescu, MD, Principal Investigator — Tameside & Glossop Integrated Care NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Tameside General Hospital, Ashton-under-Lyne
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: No